CLINICAL TRIAL: NCT05408026
Title: A Phase II, Multicenter, Open-Label Study of the Combination of Pomalidomide, Bortezomib, Low-Dose Dexamethasone, and Daratumumab in Patients With Relapsed or Refractory Multiple Myeloma
Brief Title: Study of Combination POM, BTZ, Low-Dose DEX, and DARA (PVD-DARA) in Patients With RRMM
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study withdrawn, trial therapy deemed no longer novel and there was a lack of site interest.
Sponsor: Alliance Foundation Trials, LLC. (Other)
Collaborators: Janssen, LP (Industry); Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AFT-35
Record Dates: First submitted 2022-05-06; First posted 2022-06-07 (Actual); Last update posted 2023-01-27 (Actual); Status verified 2023-01

CONDITIONS: Relapsed or Refractory Multiple Myeloma
MeSH Terms: conditions — Recurrence; Multiple Myeloma | interventions — daratumumab; Dexamethasone; pomalidomide; Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Combination of Pomalidomide, Bortezomib, Low-Dose Dexamethasone, and Daratumumab (Experimental): Combination of Pomalidomide, Bortezomib, Low-Dose Dexamethasone, and Daratumumab
  Interventions: Drug: Daratumumab; Drug: Pomalidomide

INTERVENTIONS:
Drug: Daratumumab — Daratumumab (and hyaluronidase) will be given over 3-5 minutes subcutaneously (under the skin) in the clinic at alternating left/right abdominal sites. Patient will take dexamethasone orally (by mouth) either before coming to clinic or in clinic, before other medications.
  Only for the first cycle, patient will receive on Day 1 daratumumab (which is mixed with a compound called hyaluronidase) and dexamethasone, 1 day before patient start the other 2 medications.
  Other Names: Dexamethasone
Drug: Pomalidomide — On day 2 of cycle 1, patient will start the other medications and will therefore receive bortezomib administered subcutaneously (SC) over 3-5 minutes and dexamethasone given orally (by mouth), either before coming to clinic or in clinic, before bortezomib. Patient will also start pomalidomide on the same day, which patient will take that evening at home and every evening for 21 days.
  Other Names: Bortezomib

SUMMARY:
This phase II clinical trial design with a safety run-in period will be used to assess the rate of VGPR or better for the combination PVD-Dara in the treatment of RRMM.

DETAILED DESCRIPTION:
A phase II clinical trial design, including an initial safety run-In period, will be used to assess the rate of VGPR or better for the combination PVD-Dara in the treatment of relapsed or refractory multiple myeloma.

In the run-in period, a maximum of 12 patients will be enrolled onto the trial using the initially proposed regimen and then the trial will be temporarily closed to enrollment, until safety data is reviewed for these patients. Adverse events during the first cycle of treatment of the initially proposed regimen will be closely monitored. If the safety criteria have been met as defined in the protocol, then the trial will reopen to enrollment using the regimen as planned until a total of 72 patients have been enrolled. If safety criteria have not been met as per protocol, then the treatment regimen will be modified for the second cohort of 12 patients after discussion with the study team taking into consideration that if intolerability is due to neutropenia the regimen will be modified by lowering the dose of pomalidomide.

The phase II will begin once the safe doses have been determined in the Run-in period. this Phase II clinical trial was designed to assess whether this 4-agent combination yields a response rate of VGPR or better in more than 65% of patients.

For the regimen found tolerable in the safety period, a two-stage Phase II clinical trial design was chosen to assess whether the VGPR or better response rate is at most 50% against the alternative that the VGPR or better response rate is at least 65%.

ELIGIBILITY:
Key Inclusion Criteria:

1. Histologically confirmed diagnosis of symptomatic multiple myeloma.
2. Evidence of disease progression or refractoriness to 1 to 3 prior lines of therapy by IMWG standard criteria.
3. Prior exposure to lenalidomide and a proteasome inhibitor is mandatory.
4. Daratumumab naïve patients or Daratumumab exposed patients who are not refractory to weekly or bi-weekly daratumumab.
5. Measurable disease:

   * Serum M protein ≥ 0.5 g/dL
   * Urine M protein ≥ 200 mg/24 hours
   * Involved serum free light chains ≥ 10 mg/dL AND an abnormal serum free light chain ratio
6. ECOG Status 0-2 ≤ 14 days prior to registration
7. Adequate organ function including ≤ 14 days prior to registration defined as:

   * ANC ≥ 1.0 x 10^9/L. (Patients cannot have received G-CSF or GM-CSF within 1 week of screening or pegfilgrastim within 2 weeks of screening)
   * Platelets ≥ 75 x 10^9/L
   * Calculated Creatinine Clearance ≥ 30 mL/min
   * Total Bilirubin ≤ 1.5 x ULN except for patients with a history of elevated total bilirubin, such as in Gilbert's
   * AST, AP, ALT ≤ 3 x ULN
   * Hepatic Child-Pugh score at worse A (eligible for the phase 2 part but not for the Run-in-Period).
8. Adequate cardiac function within 8 weeks prior to registration defined as LVEF ≥ 40%.

Key Exclusion Criteria:

1. Disease refractory to weekly or bi-weekly daratumumab therapy.
2. Female patients who are lactating or have a positive serum pregnancy test ≤ 14 days from registration during the screening period.
3. Failure to have fully recovered from the reversible effects of prior anti-cancer therapy.
4. Major surgery within 14 days before registration.
5. Focal radiation therapy within 14 days prior to randomization with the exception of palliative radiotherapy for symptomatic management but not on measurable extramedullary plasmacytoma.
6. Disease-related central nervous system involvement.
7. Plasma cell leukemia, AL amyloidosis, or POEMS syndrome.
8. The subject has uncontrolled significant intercurrent illness including, but not limited to, ongoing or active infection, uncontrolled congestive heart failure, New York Heart Association Class III-IV, unstable angina pectoris, stroke, myocardial infarction, uncontrolled cardiac arrhythmias < 6 months prior to registration, or uncontrolled hypertension.
9. Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol.
10. Known allergy to any of the study medications, their analogues, or excipients in the various formulations of any agent.
11. Known GI disease or GI procedure that could interfere with the oral absorption of study medication including difficulty swallowing.
12. Concurrent malignancy except for treated non-melanoma skin cancer, cervical carcinoma in situ and low-risk prostate CA being monitored without treatment.
13. Grade 2 and higher peripheral neuropathy on clinical examination ≤ 14 days prior to registration.
14. Chemotherapy ≤ 14 days prior to registration.
15. Exposure to an investigational drug (including investigational vaccine) or invasive investigational medical device for any indication within 4 weeks or 5 pharmacokinetic half-lives, whichever is longer.
16. Patients with known chronic obstructive pulmonary disease (COPD) with a forced expiratory volume in 1 second (FEV1) <50% of predicted normal; moderate or severe persistent asthma within the past 2 years, or uncontrolled asthma of any classification. Note.
17. Moderate or severe persistent asthma within the past 2 years, or uncontrolled asthma of any classification. Note that participants who currently have controlled intermittent asthma or controlled mild persistent asthma are allowed to participate.
18. Patients who have a contraindication to the use of any form of anticoagulation or antiplatelet agents.
19. Patient who are on a strong CYP34A or CYP1A2 inducer or inhibitors
20. Patients with Hepatic Child-Pugh score B and C. Note that Hepatic Child-Pugh score A are excluded from the Run-in-Period of the trial
21. Patient is:

    * seropositive for human immunodeficiency virus (HIV).
    * seropositive for hepatitis B (defined by a positive test for hepatitis B surface antigen [HBsAg]). Subjects with resolved infection (ie, subjects who are HBsAg negative but positive for antibodies to hepatitis B core antigen [anti-HBc] and/or antibodies to hepatitis B surface antigen [anti-HBs]) must be screened using real-time polymerase chain reaction (PCR) measurement of hepatitis B virus (HBV) DNA levels. Those who are PCR positive will be excluded. EXCEPTION: Subjects with serologic findings suggestive of HBV vaccination (anti-HBs positivity as the only serologic marker) AND a known history of prior HBV vaccination, do not need to be tested for HBV DNA by PCR.
    * seropositive for hepatitis C (except in the setting of a sustained virologic response [SVR], defined as aviremia at least 12 weeks after completion of antiviral therapy).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Safety Run-In Stage: Adverse events (AEs) will be assigned a grade and attribution using CTCAE v5.0 to determine the presence of dose-limiting toxicities (DLT). | 4-9 months
  DLTs will be used to assess the safety profile & determine tolerability of PVD-DARA in patients with RRMM. A DLT is the occurrence of any below toxicity during the first cycle probably, possibly or definitely related to study treatment:
  * Grade 4 neutropenia
  * Febrile neutropenia
  * Grade 4 thrombocytopenia
  * Grade 3 thrombocytopenia w/ bleeding
  * Grade 4 anemia, unexplained by underlying disease
  * Any non-hematological toxicity Grade ≥ 3, except:
    * Alopecia
    * Grade 3 nausea/vomiting/diarrhea for < 72 hours w/ antiemetic & other supportive care
    * Grade 3 fatigue for < 1 week
    * Grade ≥ 3 isolated electrolyte abnormalities for ≤ 72 hours, not clinically complicated, resolve spontaneously/respond to conventional medical interventions
    * Grade ≥ 3 amylase/lipase elevation not associated w/ symptoms/clinical manifestations of pancreatitis
    * Grade 3 tumor lysis syndrome for ≤ 72 hours, not clinically complicated, resolves spontaneously/responds to conventional medical intervention
Phase II: To estimate the rate of Very Good Partial Response (VGPR) or better after 8 cycles of the combination PVD-DARA in patients with RRMM, including those with prior exposure to daratumumab | 36 months
  To estimate the rate of VGPR or better after 8 cycles of the combination PVD-DARA in patients with RRMM, including those with prior exposure to daratumumab

SECONDARY OUTCOMES:
Rate of Adverse Events Grade ≥ 3 [Toxicity Profile] | 4 years
  The toxicity profile will be summarized by determining the rate of patients with a grade 3 or higher adverse event.
Rate of Dose Omission [Toxicity Profile] | 4 years
  The toxicity profile will be summarized by determining the rate of patients at least one omitted dose.
Rate of Dose Modification [Toxicity Profile] | 4 years
  The toxicity profile will be summarized by determining the rate of patients at least one modified dose.
To determine the overall response rate (ORR, including sCR, CR, VGPR, PR) after 8 cycles of the combination PVD-DARA in patients with RRMM, including patients previously exposed to daratumumab | 4 years
  To determine the overall response rate (ORR, including sCR, CR, VGPR, PR) after 8 cycles of the combination PVD-DARA in patients with RRMM, including patients previously exposed to daratumumab
To determine the Progression Free Survival (PFS) for the combination PVD-DARA in patients with RRMM, including patients previously exposed to daratumumab | 4 years
  To determine the Progression Free Survival (PFS) for the combination PVD-DARA in patients with RRMM, including patients previously exposed to daratumumab
To determine the overall survival for the combination PVD-DARA in patients with RRMM, including patients previously exposed to daratumumab | 4 years
  To determine the overall survival for the combination PVD-DARA in patients with RRMM, including patients previously exposed to daratumumab

IPD SHARING:
Plan to Share IPD: No